CLINICAL TRIAL: NCT06164392
Title: Evaluation of Neuroma Perfusion with Indocyanine Green Fluorescence Angiography
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The attendings who were to participate did not want to alter their standard neuroma treatment of neurotomy and TMR, as opposed to dissecting the end of all neuromas before neurotomy. No patients were enrolled in the study.
Sponsor: Northwestern University (Other)
Collaborators: American Society for Surgery of the Hand (Other)
Responsible Party: Principal Investigator, Gregory A Dumanian, Chief of Plastic surgery in the Department of Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00220008
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Neuroma; Neuroma Amputation; Neuroma of Upper Limb; Neuroma of Lower Limb
Keywords: Neuroma; Indocyanine Green; Targeted Muscle Reinnervation; Regenerative Peripheral Nerve Interface; Nerve Repair; Fluorescence Angiography
MeSH Terms: conditions — Neuroma | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neuroma ICG (Experimental): Subjects will receive Intravenous ICG to generate a Fluorescence Angiogram of the Neuroma
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Intravenous administration of indocyanine green followed by fluorescence angiography imaging of the neuroma
  Other Names: ICG

SUMMARY:
The purpose of this study is to characterize the perfusion of neuromas using indocyanine green fluorescence angiography

DETAILED DESCRIPTION:
Neuromas represent the frustrated regeneration of injured nerve axons encased in a bulbous scar. Symptomatic neuromas are particularly problematic in patients with amputations. Targeted Muscle Reinnervation is a novel surgical approach to neuroma treatment, resulting in improved residual limb pain in amputees. Nevertheless, a subset of Targeted Muscle Reinnervation patients achieve inadequate relief. Incomplete neuroma excision may be of particular concern in such cases, as failure to completely excise the neuroma risks leaving a scarred proximal nerve stump behind. Despite the critical importance of complete neuroma excision, there is no clear definition of a neuroma's "zone of injury". Indeed, intraoperatively determining where to cut a nerve to ensure accurate and complete excision of a neuroma at the time of reconstruction or repair is an unsolved problem in peripheral nerve surgery. The proposed research aims to characterize the perfusion of neuromas using fluorescence angiography. Specifically, we will test the hypothesis that intravascular indocyanine green (ICG) renders visible the perturbations in nerve perfusion associated with neuromas, and that these altered perfusion patterns correlate with the nerve's "zone of injury" as identified by histopathology. Ultimately, indocyanine green (ICG) fluorescence angiography may facilitate intraoperative decision-making at the time of neuroma excision.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical diagnosis of neuroma
* Scheduled elective surgery for neuroma excision

Exclusion Criteria:

* Minors, or age < 18 years old at the time of surgery
* Unable to provide written, informed consent
* Prisoners and decision-impaired individuals
* Pregnant or lactating women
* History of allergy to indocyanine green
* History of allergy to iodides
* History of allergic asthma
* History of hepatic failure
* History of renal failure
* Patients in whom the planned surgical incision/approach does not include excision of the neuroma
* Patients in whom adequate surgical exposure of the neuroma is unable to be obtained, as determined intraoperatively at the time of surgery by the Investigator or Co-Investigators
* Any subject who, at the discretion of the Investigator or Co-Investigators, is not suitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-28 (Estimated); Primary Completion 2024-12-28 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Neuroma ICG Fluorescence Angiogram | Intraoperative
  Nerve Tissue Perfusion as visualized by Fluorescence Angiogram

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Dumanian, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: For one year following publication
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact gdumania@nm.org